CLINICAL TRIAL: NCT04570540
Title: Obesity in Sleep Medicine - Focusing on OHS Phenotypes
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor
Other Study IDs: WI_137/2013
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
Keywords: Obstructive Sleep Apnea; Sleep Hypoventilation
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Sleep Apnea, Obstructive | interventions — Polysomnography; Respiratory Function Tests; Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OSA: Obstructive Sleep Apnea as confirmed by full-night attended in-lab polysomnography showing an apnea-hypopnea index of >=15 per hour or, alternatively, an apnea-hypopnea index >=5 with excessive daytime sleepiness as defined by an Epworth Sleepiness Scale score >9.
  Interventions: Diagnostic Test: Sleep Study; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Hypercapnic ventilatory response; Diagnostic Test: Cardiopulmonary Exercise Test
- OSA+SH: Obstructive Sleep Apnea as confirmed by full-night attended in-lab polysomnography showing an apnea-hypopnea index of >=15 per hour or, alternatively, an apnea-hypopnea index >=5 with excessive daytime sleepiness as defined by an Epworth Sleepiness Scale score >9. Furthermore, co-existing hypoventilation during sleep, defined by the presence of intermittent hypercapnia as measured by transcutaneous capnometry and arterialized capillary blood gas analysis.
  Interventions: Diagnostic Test: Sleep Study; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Hypercapnic ventilatory response; Diagnostic Test: Cardiopulmonary Exercise Test
- OHS: Obstructive Sleep Apnea as confirmed by full-night attended in-lab polysomnography showing an apnea-hypopnea index of >=15 per hour or, alternatively, an apnea-hypopnea index >=5 with excessive daytime sleepiness as defined by an Epworth Sleepiness Scale score >9. Furthermore, co-existing hypoventilation during wakefulness, defined by a PCO2>45mmHg as measured by arterialized capillary blood gas analysis.
  Interventions: Diagnostic Test: Sleep Study; Diagnostic Test: Pulmonary Function Test; Diagnostic Test: Hypercapnic ventilatory response; Diagnostic Test: Cardiopulmonary Exercise Test

INTERVENTIONS:
Diagnostic Test: Sleep Study — Full-night attended in-lab polysomnography with accompanying transcutaneous capnometry
Diagnostic Test: Pulmonary Function Test — Bodyplethysmographic assessment
Diagnostic Test: Hypercapnic ventilatory response — Measurement of hypercapnic ventilatory response based on the method described by Read in 1967, using a rebreathing bag
Diagnostic Test: Cardiopulmonary Exercise Test — Symptom-limited cardiopulmonary exercise test with a ramp protocol according to the ATS/ACCP and ERS recommendations

SUMMARY:
This study focuses on a comprehensive examination of obese patients with sleep-related breathing disorders including patients with OSA, sleep hypoventilation and OHS. The aim of this study is to (1) evaluate characteristics of and differences between severity levels of obesity-related breathing disorders, (2) discuss pathophysiological variables associated with hypoventilation during sleep or at daytime and (3) find functional parameters indicating sleep hypoventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* BMI ≥ 30 kg/m²
* Indication for sleep lab admission or indication for BiLevel or non-invasive ventilation therapy initiation due to existing hypoventilation/OHS

Exclusion Criteria:

* Age <18 years
* Pregnancy, Lactation
* Any medical, psychological or other condition impairing the patient's ability to provide informed consent.
* Missing informed consent
* Participation in another clinical study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obese patient routinely admitted to sleep lab
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-04-24 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Hypercapnic ventilatory response | Within 48 hours of sleep lab admission

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Chief Physician
Locations (1):
- Institut für Pneumologie an der Universität zu Köln / Wissenschaftliches Institut Bethanien für Pneumologie e.V., Solingen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herkenrath SD, Treml M, Hagmeyer L, Matthes S, Randerath WJ. Severity stages of obesity-related breathing disorders - a cross-sectional cohort study. Sleep Med. 2022 Feb;90:9-16. doi: 10.1016/j.sleep.2021.12.015. Epub 2022 Jan 4. PMID 35051737